CLINICAL TRIAL: NCT05281731
Title: Sonobiopsy for Noninvasive and Sensitive Detection of Glioblastoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202202025; R01CA276174 (NIH)
Record Dates: First submitted 2022-02-11; First posted 2022-03-16 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Sonobiopsy (Experimental): * Once enrolled, participants would be prepared for standard of care surgery.
  * The sonobiopsy involves the standard procedure for a biopsy, but the biopsy needle is replaced with a customized ultrasound probe, a standard ultrasound contrast agent (microbubbles) is injected intravenously, and the probe is turned on for 3 minutes for the sonobiopsy. Then the planned surgery to remove the tumor will occur.
  * An additional brief MRI scan will be obtained using the intraoperative MRI to define imaging changes (if any) that occur as a result of the sonobiopsy procedure. The imaging protocols will include a 3D T2-weighted (T2w) scan, and 3D contrast T1-weighted (T1w) with dynamic contrast enhancement and if time allows T2* sequence.
  * Blood will be collected at several time points.
  * A small skin biopsy or another blood draw will be drawn for comparison against the genetic mutations shown in the tumor.
  * The blood, tumor, and skin (if applicable) will undergo genetic analysis.
  Interventions: Device: Sonobiopsy; Procedure: Research blood; Genetic: Cancer Personalized Profiling; Device: Definity®

INTERVENTIONS:
Device: Sonobiopsy — Ultrasound combined with microbubbles to facilitate sampling of biomarkers from brain tumors via blood-based liquid biopsy
Procedure: Research blood — No more than 10 minutes prior to ultrasound sonication, 10 minutes after ultrasound sonication, 30 minutes after ultrasound sonication (optional at the discretion of the PI), and 60 minutes after ultrasound sonication (optional at the discretion of the PI)
Genetic: Cancer Personalized Profiling — Cancer Personalized Profiling by deep Sequencing will be used to compare the frequency of tumor-specific variants in the blood before and after sonobiopsy.
Device: Definity® — Being used off-label in this trial
  Other Names: Definity® microbubbles

SUMMARY:
This clinical study to evaluate sonobiopsy is significant because sonobiopsy will fundamentally enhance the clinician's insight into the molecular features of an intracranial lesion to tailor treatment approaches and optimize outcomes. In addition to the standard diagnostics of anatomic imaging and surgical histology, sonobiopsy has the potential to become the third pillar for brain tumor management by radically advancing the ability to easily and regularly acquire tumor genetic and molecular signatures. This enhanced capability will have a dramatic impact on patient survival and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Must be newly diagnosed with a lesion in the brain with imaging characteristics consistent with glioblastoma multiforme. Scan must have occurred no more than 28 days prior to enrollment.
* Lesion must be > 3 cm in maximal dimension on MRI.
* Lesion must be in the supratentorial space within 5 cm of the cortical surface.
* Lesion must be gadolinium enhancing.
* Low grade tumors and metastatic tumors
* Recurrent brain tumors and/or radiation necrosis
* Must be planning to undergo surgical resection of the tumor.
* Must be at least 18 years old.
* Patients with recurrent GBM who are planning to undergo surgical resection or laser ablation of the recurrent tumor. Recurrence must be confirmed on MRI performed no more than 28 days prior to enrollment.

Exclusion Criteria:

* Contraindication to MRI.
* Previous cranial surgery.
* Previous history of cancer and/or cancer treatments.
* Coagulopathy within 14 days of enrollment defined as PT/PTT outside of normal parameters and platelets < 100,000/mcL.
* Physical skull defect of any kind.
* Ferrous material in the scalp or skull.
* Scalp or skin disease that limits contact with the ultrasound probe.
* Enrolled in another clinical trial where intervention is administered prior to surgery.
* Known hypersensitivity to polyethylene glycol.
* Known unstable cardiopulmonary condition (e.g. acute myocardial infarction, acute coronary artery syndromes, worsening or unstable congestive heart failure, serious ventricular arrhythmias).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of sonobiopsy as measured by change in ctDNA level | Day 1
  The feasibility of sonobiopsy will be demonstrated by an increase in the amount of ctDNA in the blood samples acquired post than prior sonobiopsy in at least 50% of the patients.
Number of matched mutations between the post-sonobiopsy sample and the tumor tissue sample | Day 1
  The agreement of the post-sonobiopsy sample mutation detected in the blood with a variant identified in the tumor tissue will be compared using a kappa statistic.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Kim, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu